CLINICAL TRIAL: NCT02956707
Title: Impact of Pre-operative Steroids on Adrenal Insufficiency and Clinical Outcomes After Neonatal Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Impact of Pre-operative Steroids on Adrenal Insufficiency
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Santiago Borasino, MD, Interim Director Pediatric Cardiac Critical Care, University of Alabama at Birmingham
Other Study IDs: F160616001
Record Dates: First submitted 2016-10-14; First posted 2016-11-07 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Adrenal Insufficiency Neonatal
Keywords: neonates; cardiopulmonary bypass; adrenal insufficiency; congenital heart disease
MeSH Terms: conditions — Adrenal Insufficiency; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — As a separate portion to this study consenting subject's legally authorized representative can provide consent to allow specimens to be stored for future research related to heart disease. These specimens include: blood (cell pellet and plasma), urine, and peritoneal dialysis fluid (if applicable).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No pre-operative steroids: This is a prospectively enrolling group of 40 subjects.
  Our current clinical practice has changed. We no longer administer pre-oeprative steroids to neonates undergoing surgery with cardiopulmonary bypass. These patients still receive their post-operative steroid infusion that starts after termination from bypass. This is their standard of care and does not change due to study enrollment.
  Subject's enrolled in this trial have a ACTH stimulation test performed: pre-operative, immediately post-cardiopulmonary bypass prior to the initiation of their clinical steroids, and prior to leaving the cardiac intensive care unit.
  Interventions: Other: No pre-operative steroids
- Pre-operative steroids: This is a retrospective group of 40 subjects who were previously administered pre-operative steroids. These subjects also had ACTH testing performed pre-operative and immediately post-separation from cardiopulmonary bypass.

INTERVENTIONS:
Other: No pre-operative steroids — Due to new information provide from previous studies at our center the investigator instituted a clinical practice change remove steroid administration in the pre-operative period for all neonates undergoing surgery with cardiopulmonary bypass. This study is to evaluate this change.
  Groups: No pre-operative steroids

SUMMARY:
Little is known regarding the incidence and clinical impact of AI in neonates during the acute postoperative period following separation from CPB. In a randomized control pilot study performed by the UAB CVICU research team, prophylactic post-CPB hydrocortisone infusions improved some postoperative outcomes, especially in those that acquired AI7. In an attempt to further explore post-CPB AI, a retrospective analysis of data from this study was performed. Of the 40 neonates included in the study, one-third (32.5%) developed AI following CPB (as determined by low-dose, 1 µg, cosyntropin stimulation test). Almost all of these subjects had normal response to cosyntropin stimulation pre-CPB. Subjects that developed AI demonstrated more hemodynamic instability, increased serum lactate and required more colloid resuscitation in the immediate post-CPB period in the operating room. Recent evidence has begun to highlight potential morbidity associated with perioperative steroid administration. Our cardiac surgery program is changing clinical practice and ceasing to give preoperative steroids to all patients (previously only neonatal CPB patients received preoperative methylprednisolone). With the possibility that preoperative steroid administration, and not CPB, primarily causes the high incidence of AI, it is prudent to further investigate the benefit and/or harm of perioperative steroid administration

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) induces systemic inflammatory response syndrome (SIRS), which may contribute to postoperative morbidity. Neonates experience an exaggerated inflammatory response and may be at a higher risk for the deleterious effects of CPB. SIRS may disrupt the hypothalamic-pituitary-adrenal (HPA) axis leading to a relative adrenal insufficiency (AI) after neonatal CPB. There is some emerging evidence supporting an association of AI with morbidity in neonates after cardiac surgery. Postoperative steroids may offer hemodynamic benefits to neonates suffering from low cardiac output syndrome (LCOS) following CPB. Benefit of postoperative steroids is multifactorial including: suppression of inflammatory cytokines, direct actions on the heart and vascular smooth muscle, and treatment of AI in a subset of patients.

Little is known regarding the incidence and clinical impact of AI in neonates during the acute postoperative period following separation from CPB. In a randomized control pilot study performed by the UAB CVICU research team, prophylactic post-CPB hydrocortisone infusions improved some postoperative outcomes, especially in those that acquired AI. In an attempt to further explore post-CPB AI, a retrospective analysis of data from this study was performed. Of the 40 neonates included in the study, one-third (32.5%) developed AI following CPB (as determined by low-dose, 1 µg, cosyntropin stimulation test). Almost all of these subjects had normal response to cosyntropin stimulation pre-CPB. Subjects that developed AI demonstrated more hemodynamic instability, increased serum lactate and required more colloid resuscitation in the immediate post-CPB period in the operating room.

In this retrospective analysis by Crawford et al.8 ACTH levels were found to be significantly lower post-CPB compared to preoperative levels. This may be secondary to a blunted HPA axis caused by preoperative methylprednisolone (all patients received), which could result in transient, iatrogenic AI. Serum cytokines were not significantly different in patients exhibiting AI compared to those with a normal adrenal response indicating that increased inflammation was not primarily responsible for the development of AI. Higher methylprednisolone levels result in higher cortisol levels due to cross-reactivity of the assays; patients with higher baseline postoperative cortisol levels demonstrated a blunted response to cosyntropin suggesting that these patients may have higher blood concentrations of methylprednisolone and its metabolites, thereby leading to more inhibition of the HPA axis. Taken together, these two studies demonstrate that AI occurs at high frequency after neonatal CPB and that AI is associated with deleterious outcomes. While postoperative hydrocortisone improves outcomes in neonates with AI, the investigator cannot exclude preoperative methylprednisolone as a cause of iatrogenic AI. Other investigators have shown in children treated with dexamethasone prior to surgery, that higher measured levels of dexamethasone were associated with postoperative AI9.

The majority of congenital heart surgery centers utilize perioperative steroids in neonates undergoing cardiac surgery with the rationale that it modulates post-CPB SIRS and treats/prevents AI; studies have inconsistently demonstrated benefit of this approach. Additionally, recent evidence has begun to highlight potential morbidity associated with perioperative steroid administration. Our cardiac surgery program is changing clinical practice and ceasing to give preoperative steroids to all patients (previously only neonatal CPB patients received preoperative methylprednisolone). With the possibility that preoperative steroid administration, and not CPB, primarily causes the high incidence of AI, it is prudent to further investigate the benefit and/or harm of perioperative steroid administration.

With these facts in mind, the investigator designed this study to determine the impact of preoperative steroid administration on development of AI and other outcomes after neonatal cardiac surgery.

B. Herein the investigator proposes to test the following HYPOTHESES and address these SPECIFIC AIMS:

HYPOTHESES: Preoperative steroid (methylprednisolone) administration is associated with development of iatrogenic AI; AI leads to increased postoperative morbidity. Preoperative steroids do not have important impact on other postoperative clinical outcomes.

SPECIFIC AIM# 1: Determine the incidence of AI (as diagnosed by 1µg cosyntropin stimulation testing) following CPB in neonates who do not receive preoperative steroids; compare to the previous cohort that received preoperative steroids.

SPECIFIC AIM# 2: Compare ACTH and cortisol levels between the two cohorts of neonates (those who do and those who do not receive preoperative steroids).

SPECIFIC AIM# 3: Compare secondary clinical outcomes including volume of crystalloid/colloid administered in the CVOR, hemodynamic parameters, laboratory values, vasoactive-inotrope score (VIS), duration of mechanical ventilation, fluid overload and mortality of the two cohorts of neonates.

ELIGIBILITY:
Inclusion Criteria:40 consecutive neonates (≤30 days of age) with complex congenital heart disease undergoing cardiac surgery with CPB who will not be given preoperative steroids.

- Controls: 40 neonates with complex congenital heart disease undergoing cardiac surgery with CPB who received two doses of preoperative methylprednisolone (10mg/kg at eight hours and one hour prior to their operation). Data from this cohort has already been prospectively collected during the original pilot randomized control trial. Based on our clinical data over the past 8 years, the demographic and risk factors of the two cohorts will be very similar.

Exclusion Criteria: Neonates who do not require CPB during cardiac surgery or fail to separate from CPB in the operating room.

-

Ages: 1 Day to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates less than 30 days old undergoing cardiac surgery with cardiopulmonary bypass who do not receive pre-operative steroid administration as part of their standard of care medical management.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
Incidence of AI in neonates who do not receive preoperative methylprednisolone | 1 year

SECONDARY OUTCOMES:
Hemodynamic parameters-Heart rate | 1.5 hours post-CPB
  hemodynamic parameters collected every 15 minutes post-CPB for 1.5 hours or until the end of the procedure-heart rate
Hemodynamic parameters- Blood pressure | 1.5 hours post-CPB
  hemodynamic parameters collected every 15 minutes post-CPB for 1.5 hours or until the end of the procedure systolic blood pressure
Hemodynamic parameters- Central venous pressure | 1.5 hours post-CPB
  hemodynamic parameters collected every 15 minutes post-CPB for 1.5 hours or until the end of the procedure central venous pressure
Hemodynamic parameters- Flank Near infrared spectroscopy | 1.5 hours post-CPB
  hemodynamic parameters collected every 15 minutes post-CPB for 1.5 hours or until the end of the procedure flank near infrared spectroscopy.
Hemodynamic parameters- cerebral near infrared spectroscopy | 1.5 hours post-CPB
  hemodynamic parameters collected every 15 minutes post-CPB for 1.5 hours or until the end of the procedure cerebral near infrared spectroscopy.
Laboratory values- lactacte | 1 week post-CPB
  serum lactate
Laboratory values- Hematocrit | 1 week post-CPB
  hematocrit
Laboratory values- hemoglobin | 1 week post-CPB
  hemoglobin
Laboratory values- Mixed venous | 1 week post-CPB
  mixed venous oxygen saturation
Laboratory values- carbon dioxide | 1 week post-CPB
  veno-arterial carbon dioxide difference is the carbon dioxide from the venous blood gas minus the carbon dioxide from the arterial blood gas.
Laboratory values- oxygen content | 1 week post-CPB
  arterial and venous oxygen content is the saturation from the arterial blood gas and the saturation from the venous blood gas
Colloid/blood product volumes administered in the cardiovascular operating room | intraoperative period
  volume in mililiters of crystalloids and colloids (albumin, fresh frozen plasma, packed red blood cells, and platelets) administered in the operating room
Inotrope infusion doses | 48 hours post-CPB
  incidence of low cardiac output syndrome based on inotropic support requirement in the post-operative period
Inflammatory cytokines | 48 hours post-CPB
  plasma will be collected and sent for inflammatory cytokine analysis at the following time points: pre-operative, 0 hour, 4 hour, 24 hour, and 48 hour post-cardiopulmonary bypass
ACTH stimulation test | 14 days post-CPB
  ACTH testing will be performed preoperative, immediately post-CPB, and prior to CICU discharge. This testing includes the following:
  Baseline ACTH and cortisol levels, administration of cosyntropin, 30 minutes post-cosyntropin cortisol level

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
On de-identified study data will be published